CLINICAL TRIAL: NCT04913701
Title: Observational Study for SARS-Cov2 Epidemiological Surveillance on Healthcare Workers and Patients in a Rehabilitation Medicine Facility
Brief Title: COVID-19 Epidemiological Surveillance on Healthcare Workers and Patients in a Rehabilitation Medicine Facility
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 20/09 main
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: SARS-Cov2
Keywords: SARS-Cov2; Covid-19; Epidemiological surveillance; Observational study; Healtcare workers; Real-life; Rehabilitation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1 - Health workers: A total number of 200-300 healthcare workers, exposed to close contact with patients, will be asked to participate to the study and will be asked to sign the informed consent.
  Interventions: Other: Observation group 1
- 2 - Patients: A total number of 100-200 patients admitted to the rehabilitation facility, referred from other healthcare facilities or from their own home, will be asked to participate to the study.
  Interventions: Other: Observation group 1
- 3 - Real life participants: A total number of 100 real-life participants, will be represented by volunteers (other employees, staff not in contact with patients
  Interventions: Other: Observation group 1

INTERVENTIONS:
Other: Observation group 1 — Subjects will be followed with 3 swabs and serological test

SUMMARY:
The recent SARS-CoV2 pandemic has highlighted that the transmission of the virus within health care facilities plays a fundamental role in its propagation and, therefore, in the increase in COVID-19 cases registered among patients and healthcare workers.

This study, original for the current lack of data on nosocomial transmission mechanisms compared to what happens in the community, proposes to conduct a study in patients, health workers and people in real-life setting.

The study will be monocentric and performed at the San Raffaele Pisana Institute in Rome, that is able to guarantee the necessary number and the right case-mix that will allow to evaluate any possible correlations between infection and pre-existing disease.

DETAILED DESCRIPTION:
Furthermore, hospitals, especially those dedicated to chronic patients, as well as other communities that are not completely closed (such as school and work communities), are also at greater risk of small outbreaks that also affect healthcare professionals.

It is therefore necessary to carry out periodic checks on all healthcare professionals who work in healthcare facilities both to ensure their health and avoid the risk of possible contamination and to prevent the possible transmission of infection from the community to the hospital.

Another essential aspect to prevent infection in such facilities is the control of colonization in admitted patients.

Negativity from SARS-CoV2 should be carefully monitored in these patients prior to their placement in different departments.

On this basis, the study aims to determine the presence of SARS-CoV2 by monitoring with serial nasopharyngeal swabs carried out on healthcare professionals working within the facility and on new patients admitted.

In order to exclude the possibility of false negatives due to low viral load found in the early stages of infection (incubation time) or any exposure that may occur in the days following the execution of the swab, the study will i provide for the repetition of the swab examination, 3 times, at weekly intervals.

In order to verify the correspondence between the presence of IgM and IgG antibodies against the virus and the positivity to the swabs, the healthcare professionals and patients who undergoing nasopharyngeal swab will be previously subjected to the rapid antibody detection test (prick test for IgG and IgM).

ELIGIBILITY:
Inclusion Criteria:

* Patients/Participants > 18 years
* Subjects who agree with the study signing the informed consent

Exclusion Criteria:

* Age <18 years;
* Pregnancy in progress;
* Simultaneous participation in another clinical study
* Ongoing immunosuppressive therapy or during the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study will be on healthcare workers in direct contact with patients (pts). Surveillance will be done on new admitted pts to evaluate prevalence of infection among pts in pulmonary, or cardiac rehabilitation.
  Data will allow to reconstruct eventual transmission and compare values observed in healthcare and real life. Random samples will be done in subjects from the population without obvious risk factors.
  Study will have 3 groups:
  * 200-300 healthcare workers in direct patients contact, incl. staff at registration desk. 100-200 pts admitted to rehabilitation at the Institute, referred from other health facilities will be enrolled in the study.
  * 100 volunteers in Real-life will be other employees, staff not in contact with patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with positive RT-PCR against SARS-CoV2 | 15 days
  All subjects will have 3 swabs done and analyzed

SECONDARY OUTCOMES:
Number of participants with qualitative IgM/IgG positive results | 15 days
  All subjects will have 1 blood pick-test

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Tomino, PhD, Study Director — IRCCS San Raffaele Pisana
Locations (1):
- IRCCS San Raffaele Pisana, Rome, Italy

REFERENCES:
- [Background] Gao WJ, Li LM. [Advances on presymptomatic or asymptomatic carrier transmission of COVID-19]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Apr 10;41(4):485-488. doi: 10.3760/cma.j.cn112338-20200228-00207. Chinese. PMID 32141279
- [Background] Gates B. Responding to Covid-19 - A Once-in-a-Century Pandemic? N Engl J Med. 2020 Apr 30;382(18):1677-1679. doi: 10.1056/NEJMp2003762. Epub 2020 Feb 28. No abstract available. PMID 32109012
- [Background] Heymann DL. Data sharing and outbreaks: best practice exemplified. Lancet. 2020 Feb 15;395(10223):469-470. doi: 10.1016/S0140-6736(20)30184-7. Epub 2020 Jan 24. No abstract available. PMID 31986258
- [Background] Hellewell J, Abbott S, Gimma A, Bosse NI, Jarvis CI, Russell TW, Munday JD, Kucharski AJ, Edmunds WJ; Centre for the Mathematical Modelling of Infectious Diseases COVID-19 Working Group; Funk S, Eggo RM. Feasibility of controlling COVID-19 outbreaks by isolation of cases and contacts. Lancet Glob Health. 2020 Apr;8(4):e488-e496. doi: 10.1016/S2214-109X(20)30074-7. Epub 2020 Feb 28. PMID 32119825
- [Background] Huh S. How to train health personnel to protect themselves from SARS-CoV-2 (novel coronavirus) infection when caring for a patient or suspected case. J Educ Eval Health Prof. 2020 Jan;17:10. doi: 10.3352/jeehp.2020.17.10. Epub 2020 Mar 7. No abstract available. PMID 32150796
- [Background] Jones DS. History in a Crisis - Lessons for Covid-19. N Engl J Med. 2020 Apr 30;382(18):1681-1683. doi: 10.1056/NEJMp2004361. Epub 2020 Mar 12. No abstract available. PMID 32163699
- [Background] Lipsitch M, Swerdlow DL, Finelli L. Defining the Epidemiology of Covid-19 - Studies Needed. N Engl J Med. 2020 Mar 26;382(13):1194-1196. doi: 10.1056/NEJMp2002125. Epub 2020 Feb 19. No abstract available. PMID 32074416
- [Background] Rothe C, Schunk M, Sothmann P, Bretzel G, Froeschl G, Wallrauch C, Zimmer T, Thiel V, Janke C, Guggemos W, Seilmaier M, Drosten C, Vollmar P, Zwirglmaier K, Zange S, Wolfel R, Hoelscher M. Transmission of 2019-nCoV Infection from an Asymptomatic Contact in Germany. N Engl J Med. 2020 Mar 5;382(10):970-971. doi: 10.1056/NEJMc2001468. Epub 2020 Jan 30. No abstract available. PMID 32003551
- [Background] Reusken CBEM, Broberg EK, Haagmans B, Meijer A, Corman VM, Papa A, Charrel R, Drosten C, Koopmans M, Leitmeyer K; EVD-LabNet and ERLI-Net. Laboratory readiness and response for novel coronavirus (2019-nCoV) in expert laboratories in 30 EU/EEA countries, January 2020. Euro Surveill. 2020 Feb;25(6):2000082. doi: 10.2807/1560-7917.ES.2020.25.6.2000082. Epub 2020 Feb 11. PMID 32046815
- [Background] Xiao Y, Torok ME. Taking the right measures to control COVID-19. Lancet Infect Dis. 2020 May;20(5):523-524. doi: 10.1016/S1473-3099(20)30152-3. Epub 2020 Mar 5. No abstract available. PMID 32145766
- [Background] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Background] Xu B, Kraemer MUG; Open COVID-19 Data Curation Group. Open access epidemiological data from the COVID-19 outbreak. Lancet Infect Dis. 2020 May;20(5):534. doi: 10.1016/S1473-3099(20)30119-5. Epub 2020 Feb 19. No abstract available. PMID 32087115